CLINICAL TRIAL: NCT07249957
Title: Reducing Radiation Target Volume in Radical Radiotherapy for Stage IIb Cervical Cancer: A Single-arm Exploratory Study
Brief Title: Reducing Radiation Target Volume for Stage IIb Cervical Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Director of Dept. of Gynecological Oncology Chongqing University Cancer Hospital, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0116
Record Dates: First submitted 2025-09-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Stage IIb Cervical Cancer Radical Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radical radiotherapy for IIb cervical cancer to reduce the irradiation area (Experimental)
  Interventions: Radiation: The external irradiation area only covers the entire uterus (including the primary lesion in the cervix), bilateral parametrium, and 3 cm below the cervical/vaginal lesions.

INTERVENTIONS:
Radiation: The external irradiation area only covers the entire uterus (including the primary lesion in the cervix), bilateral parametrium, and 3 cm below the cervical/vaginal lesions. — The external irradiation area only covers the entire uterus (including the primary lesion in the cervix), bilateral parametrium, and 3 cm below the cervical/vaginal lesions.

SUMMARY:
This is a domestic single-center prospective clinical trial. The study selected patients with histologically confirmed cervical squamous cell carcinoma, diagnosed as stage IIb according to the FIGO 2018 staging principle (tumor size < 4 cm). The patients first received 6 cycles of induction chemotherapy (carboplatin (AUC2) + paclitaxel (80 mg/m2), q1w), followed by concurrent chemoradiotherapy with a platinum-based regimen. The external beam radiation field only covered the entire uterus (including the primary lesion of the cervix), the bilateral parametrium, and the lesion of the cervix/vagina extending 3 cm downward. A total of 60 participants are planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participated in this study and signed the informed consent form;
2. Age range: 50 to 75 years old;
3. Patients with cervical cancer who had not undergone surgery or chemotherapy and were initially diagnosed with squamous cell carcinoma by pathological histology, and were HPV high-risk positive;
4. According to the 2018 International Federation of Gynecology and Obstetrics (FIGO) staging system, it was stage IIb (tumor size < 4 cm);
5. ECOG score: 0 to 1, with an expected survival of more than 6 months;
6. Pregnant women must undergo a pregnancy test (serum or urine) 7 days before enrollment, and the result must be negative, and they are willing to use appropriate contraceptive methods during the trial;
7. According to the investigator's judgment, there are no absolute contraindications to radiotherapy and chemotherapy or surgery, and they can comply with the trial protocol.

Exclusion Criteria:

1. Active or uncontrolled severe infections;
2. Cirrhosis, decompensated liver disease;
3. History of immunodeficiency, including HIV positive or having other acquired congenital immune deficiency diseases;
4. Chronic renal insufficiency and renal failure;
5. Patients with other malignancies that require treatment and/or newly diagnosed within 5 years;
6. Myocardial infarction, severe arrhythmia, and ≥ grade 2 congestive heart failure (NYHA classification);
7. Patients who have undergone pelvic artery embolization;
8. Patients who have received radiotherapy for pelvic malignant tumors in the past;
9. Patients who have received partial hysterectomy or radical hysterectomy in the past;
10. Patients with a history of severe allergic reaction to platinum-based chemotherapy drugs;
11. Comorbidities, requiring the use of drugs that cause significant liver and kidney damage during treatment, such as tuberculosis, etc.;
12. Patients who cannot understand the experimental content and cannot cooperate, or who refuse to sign the informed consent form;
13. Patients with serious accompanying diseases or other special conditions that seriously endanger their safety or affect their ability to complete the study.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
1."Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0" 2."Therapeutic Effect as Assessed by RECIST1.1" | 4 years

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT07249957/Prot_SAP_000.pdf